CLINICAL TRIAL: NCT00000913
Title: A Randomized Trial of Two Saquinavir-Containing Combination Treatment Regimens in Children With HIV Infection
Brief Title: A Study to Compare Two Anti-HIV Combination Therapies Each Containing Saquinavir in HIV-Positive Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 397; 11353 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Nelfinavir; Saquinavir

INTERVENTIONS:
Drug: Ritonavir
Drug: Nelfinavir mesylate
Drug: Saquinavir

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a soft-gel capsule formulation of saquinavir (SQV-SGC), a protease inhibitor, when given in combination with other anti-HIV drugs.

SQV-SGC has been tested in adults for the treatment of HIV infection, but more information is still needed about SQV-SGC in children. Recent studies suggest that this soft-gel capsule form may be safer and more effective than other protease inhibitors.

DETAILED DESCRIPTION:
Clinical trials in adults and children suggest that SQV-SGC has advantages over other protease inhibitors in terms of tolerability, safety, and effectiveness in patients who have failed therapy with other protease inhibitors. [AS PER AMENDMENT 11/24/99: Pharmacokinetic data from this study demonstrate lower than expected plasma SQV exposures, particularly in Arm 1. Based on these data, patients in the study will be offered the opportunity to adjust their doses. Ritonavir added to the Arm 1 regimen is expected to significantly increase SQV-SGC plasma levels and allow twice-daily dosing for SQV-SGC.]

Patients are randomized to one of two study arms. Patients in Arm 1 receive SQV-SGC plus two [AS PER AMENDMENT 11/24/99: one or two] NRTIs of choice. Patients in Arm 2 receive SQV-SGC plus NFV plus one or two NRTIs of choice. All participants are evaluated by physical examinations and laboratory tests during the study and are followed for incidence of death, cancer, or fetal abnormality. NRTIs are not provided as part of this study. [AS PER AMENDMENT 11/24/99: This study is closed to accrual. All subjects on follow-up (Cohort 1) are given the option of either discontinuing participation in ACTG 397 or participating in the next phase of the study (version 2.0). Those electing to continue participation constitute Cohort 1A. The adjusted Arm 1 regimen consists of SQV-SGC plus ritonavir plus one or two NRTIs. Ritonavir is not provided as part of this study. The Arm 2 regimen study drugs have not changed but the maximum allowable dose of SQV-SGC has increased from 1,200 mg twice-daily to 1,600 mg twice-daily. Participants continue to be followed with physical examinations and laboratory evaluations that include an intensive pharmacokinetics study on Day 14 of the new regimen.]

ELIGIBILITY:
Inclusion Criteria

Your child may be eligible for this study if he or she:

* Is HIV-positive.
* Is 3 to 16 years of age (consent of parent or guardian is required).
* Has an HIV level greater than 10,000 copies/ml.
* Has never taken at least one of the following anti-HIV drugs: lamivudine, zidovudine, stavudine, or didanosine.
* Is able to swallow capsules and tablets.

Exclusion Criteria

Your child will not be eligible if he or she:

* Has cancer requiring chemotherapy.
* Has an acute opportunistic (AIDS-related) infection requiring therapy.
* Has had two or more episodes of moderate or severe diarrhea or vomiting in the 3 months prior to study entry.
* Has ever taken SQV or NFV.
* Is pregnant or breast-feeding.
* Is taking certain medications, including those that would interfere with the study drugs.

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Study Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kline, Study Chair; Courtney Fletcher, Study Chair
Locations (36):
- United States (33):
  - Univ of Alabama at Birmingham / Childrens Hosp of AL, Birmingham, Alabama
  - Univ of Alabama at Birmingham - Pediatric, Birmingham, Alabama
  - Long Beach Memorial (Pediatric), Long Beach, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Children's Hosp of Oakland, Oakland, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Yale Univ Med School, New Haven, Connecticut
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami (Pediatric), Miami, Florida
  - Palm Beach County Health Dept, Riviera Beach, Florida
  - Emory Univ Hosp / Pediatrics, Atlanta, Georgia
  - Cook County Hosp, Chicago, Illinois
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Chicago Children's Memorial Hosp, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - North Shore Univ Hosp, Great Neck, New York
  - Cornell Univ Med College, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - Incarnation Children's Ctr / Columbia Presbyterian Med Ctr, New York, New York
  - Harlem Hosp Ctr, New York, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Med College of Virginia, Richmond, Virginia
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Brundage RC, Kline MW, Lindsey J, Fenton T, Fletcher CV. Pharmacokinetics of saquinavir (SQV) with nelfinavir (NFV) or ritonavir (RTV) in HIV-infected children. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 728)
- [Background] Kline MW, Fletcher CV, Lindsey JC, Fenton T. A randomized trial of two saquinavir (SQV-SGC)-containing combination treatment regimens in HIV-infected children. 7th Conference on Retroviruses and Opportunistic Infections. 2000 Jan 30-Feb 2 [Poster 694]
- [Background] Kline MW, Fletcher CV, Lindsey JC, Fenton T. A randomized trial of combination therapy with saquinavir soft gelatin capsules (SQV) in HIV-infected children. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 683)
- [Background] Brundage RC, Kline MW, Lindsey JC, Fenton T, Fletcher CV. Pharmacokinetics (PK) of saquinavir (SQV) and nelfinavir (NFV) in a twice-daily (BID) regimen in HIV-infected children. 7th Conference on Retroviruses and Opportunistic Infections. 2000 Jan 30-Feb 2 [Poster 718]